CLINICAL TRIAL: NCT00648999
Title: Phase IV, Non Randomized Study in ARV Experienced Patients Under Switch Therapy With Kaletra
Brief Title: Safety and Efficacy of Kaletra in ARV Therapy Experienced Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEXI-P01-02
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: Kaletra
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: lopinavir/ritonavir
- 2 (Active Comparator)
  Interventions: Drug: lopinavir/ritonavir

INTERVENTIONS:
Drug: lopinavir/ritonavir — lopinavir/ritonavir 400 mg/100 mg bid 48 weeks of treatment
  Other Names: ABT-378; Kaletra

SUMMARY:
To demonstrate that patients treated with Kaletra have an improvement in their quality of life compared to the quality of life they had with their previous NRTI therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infected subjects
* Subjects failing in current HIV treatment, or
* Subjects with a viral load < 400 copies/mL and not tolerating their current HIV treatment.

Exclusion Criteria:

* Subject is currently participating in another clinical study or has participated in another clinical study within 30 days prior to screening visit
* Subject is pregnant

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2003-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Baseline, Week 4, Week 24 and Week 48
CD4 | Baseline, Week 24 and Week 48

SECONDARY OUTCOMES:
Adverse Event Monitoring | Baseline, Week 4, Week 24 and Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Jose Canadas, MD, Study Director — AbbVie
Locations (13):
- Mexico (13):
  - Site Ref # / Investigator 4074, León, Guanajauto
  - Site Ref # / Investigator 4049, Mexico City, Mexico City
  - Site Ref # / Investigator 4050, Mexico City, Mexico City
  - Site Ref # / Investigator 4051, Mexico City, Mexico City
  - Site Ref # / Investigator 4077, Mexico City, Mexico City
  - Site Ref # / Investigator 4056, Mexico City, Mexico City
  - Site Ref # / Investigator 4054, Morelia, Michoacán
  - Site Ref # / Investigator 4072, Tepic, Nayarit
  - Site Ref # / Investigator 4052, Oaxaca City, Oaxaca
  - Site Ref # / Investigator 4053, Puebla City, Puebla
  - Site Ref # / Investigator 4055, Culiacán, Sinaloa
  - Site Ref # / Investigator 4075, Mérida, Yucatán
  - Site Ref # / Investigator 4073, Chihuahua City

REFERENCES:
- See also: Related Info — http://rxabbvie.com